CLINICAL TRIAL: NCT05256459
Title: Clinical Intervention Strategy for High-risk Hepatitis B Related Hepatocellular Carcinoma Based on Liquid Biopsy Screening Technique
Brief Title: Clinical Intervention Strategy for High-risk Group of Hepatitis B Related Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhang Dazhi,MD (Other)
Collaborators: Chongqing Three Gorges Central Hospital (Other); The Affiliated Hospital Of Southwest Medical University (Other); Chongqing Public Health Medical Center (Other)
Responsible Party: Sponsor-Investigator, Zhang Dazhi,MD, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: Zhangdz2017
Record Dates: First submitted 2022-01-06; First posted 2022-02-25 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group: Those who did not deal with nodules and were closely followed up.
- Treatment group: Patients with liver nodules were treated by radiofrequency ablation or/and surgery and so on.
  Interventions: Other: Long term follow-up

INTERVENTIONS:
Other: Long term follow-up — No extra intervention.
  Groups: Treatment group

SUMMARY:
This study aims to explore whether there is difference in the incidence rate and incidence rate of HCC in patients with chronic hepatitis B who are screened for high risk of liver cancer. Whether the timely intervention can be used to reduce the incidence of HCC for the early screening and early warning patients can provide evidence-based medical evidence for the selection or adjustment of anti HBV drugs in high-risk patients with liver cancer. To provide evidence for whether patients with liver nodules at high risk of liver cancer need to deal with liver nodules in advance.

DETAILED DESCRIPTION:
This study is a multicenter, prospective clinical study. Including the Second Affiliated Hospital of Chongqing Medical University, the Third Affiliated Hospital of Chongqing Medical University, the First Affiliated Hospital of Southwest Medical University, Chongqing public health treatment center and the Three Gorges central hospital.

Firstly, patients were screened for peripheral blood cfdna gene to screen patients with high risk of liver cancer. High risk patients were examined for high-precision HBV-DNA quantification, liver function, AFP, abdominal imaging (color Doppler ultrasound, CT or MR), blood map, HIV syphilis screening, anti HDV, anti HCV, etc. according to the results of high-precision HBV-DNA quantification (lower than the detection limit (< 10 IU / ml), ≥ 10 IU / ml, non negative ones are uniformly called positive), and patients are divided into 2 groups according to the wishes of patients, with 50 cases in each group. The observation group includs those who did not deal with nodules and were closely followed up，another group is treatment group，includs those who with hepatic nodules were treated by radiofrequency ablation and/or surgery and so on. Follow up examinations were conducted every 3 months to the center. The follow-up period lasted for 3 years. Clinical data were recorded, incidence rate of liver cancer, occurrence time of liver cancer and incidence of adverse events in liver were recorded.

Research implementation process and route

1. Recruitment object: after the approval of the ethics committee, the recruitment was started in each experimental center, the basic information and various examination indexes of the patients were collected, and the patients were informed that they needed to go to the outpatient clinic of our hospital for follow-up examination every 3 months, with a total follow-up of 3 years.
2. Establishment of information archives: in addition to recording the basic information and examination results of patients, it also includes the time when patients should be followed up in our hospital. Contact and inform patients in advance before each follow-up time. At the same time, special clinical events during follow-up were recorded.
3. Statistical analysis: after a three-year follow-up, the data collected by each center were tested by t-test and multivariate Cox analysis to analyze the time when patients in each group developed into primary liver cancer and the incidence of primary liver cancer in each group.
4. Data to be collected: general medical history characteristics: medical record number, name, gender, age, disease degree (whether there is decompensation / compensation of liver cirrhosis, whether there is liver nodule, etc.), enrollment time, contact information, whether to drink alcohol and medication. Examination and inspection indicators: liver function, renal function, blood chart analysis, hepatitis B two half and half, anti HCV, anti HDV, AIDS syphilis screening, high precision HBV-DNA quantification, abdominal color Doppler ultrasound (if necessary CT or MR), liver transient elastography, liver cirrhosis patients need additional coagulation. Patients undergoing radiofrequency ablation or surgical treatment of liver nodules need to record the operation time and mode.
5. Follow up: after enrollment, the relevant examination indexes were rechecked every 3 months. The follow-up period was 3 years.
6. Patients with new liver diseases and decompensated complications of liver cirrhosis also need to be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign informed consent
* Male or female, 18 ≤ age≤ 75
* The diagnosis was in accordance with the 2019 guidelines for the diagnosis and treatment of chronic hepatitis B and received anti HBV treatment for 48 weeks;
* Imaging examination showed liver nodules or space occupying lesions (any imaging examination of abdominal color Doppler ultrasound, CT and MRI), and imaging examination could not determine the benign and malignant of the lesions
* The estimated survival time is more than half a year
* Peripheral blood cfdna gene screening is high risk
* Full capacity for civil conduct

Exclusion Criteria:

* Primary liver cancer was diagnosed or supported by the following evidence: elevated alpha fetoprotein (AFP > 100ng / ml) or liver imaging showed clear liver cancer nodules in the liver
* Have a history of malignant tumors within 5 years before screening, except for specific cancers cured by surgical resection (such as basal cell skin cancer, etc.)
* Current or previous history of major diseases that may interfere with personal treatment, evaluation or compliance. Major diseases are 25 major diseases specified by the CIRC
* Combined with HCV, HIV, HDV or other infectious diseases
* Severe lung disease, severe heart disease or genetic metabolic disease
* Psychiatric hospitalization, attempted suicide and / or temporary disability due to mental illness in the past 5 years
* Combined with autoimmune liver disease, alcoholic liver disease and drug-induced liver injury
* Pregnant or lactating women
* The researcher believes that it is not suitable to participate in this experiment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hepatitis B patients who meet the inclusion conditions and do not meet the exclusion conditions。
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-10 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The patients' enrollment time. | up to 3 years.
  The time of all patients when they were enrolled.
Time the patients were diagnosed. | up to 5 years
  The time of the patients when they were diagnosed of liver cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Zhang, Doctor, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: No
There is no sharing plan